CLINICAL TRIAL: NCT03215888
Title: Effects of Change in Insulin Resistance and Systemic Inflammation After Bariatric Surgery on Brain Neurochemistry, Neuroinflammation and Cognitive Function
Brief Title: Effects of Change in Insulin Resistance and Systemic Inflammation on Brain Structure and Function
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: MED-2017-25812
Record Dates: First submitted 2017-06-30; First posted 2017-07-12 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Obesity; Bariatric Surgery Candidate
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum sample to measure hormones and inflammatory markers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese: Obese individuals undergoing bariatric surgery
  Interventions: Procedure: bariatric surgery
- controls: matched non-obese controls

INTERVENTIONS:
Procedure: bariatric surgery — Obese patients will undergo brain imaging, neurocognitive function testing and measurement of insulin resistance and inflammatory markers pre- and post bariatric surgery
  Groups: Obese

SUMMARY:
Obesity is associated with alterations in brain structure and cognitive impairment and is a risk factor for Alzheimer's disease and vascular dementia. The mechanisms underlying obesity related decline in cognitive function are not fully understood. The long-term goal of this project is to understand how obesity affects cognitive function, with the aim to develop new ways to prevent and treat obesity related cognitive decline

DETAILED DESCRIPTION:
A growing body of evidence suggests that obesity is associated with alterations in brain structure and cognitive impairment. Mid-life obesity is a risk factor for Alzheimer's disease and vascular dementia. The mechanisms underlying obesity related decline in cognitive function are not fully understood. The long-term goal of this research is to identify how obesity, insulin resistance (IR), and their treatment impact brain structure and function. The investigators propose that IR and obesity related inflammation are two modifiable factors that affect neuronal integrity and lead to cognitive dysfunction. In this proposal, investigators will test two hypotheses: 1) among obese patients planning to undergo bariatric surgery (specifically vertical sleeve gastrectomy), baseline IR and systemic and brain markers of inflammation will inversely correlate with performance on cognitive testing and correlate with abnormalities in brain structure and 2) following bariatric surgery subjects who experience the greatest reduction in IR and obesity related inflammation will have the greatest improvement in cognitive function and brain structure. To address these hypotheses, investigators will use a comprehensive battery of tests to evaluate cognition and state of the art magnetic resonance imaging (MRI) techniques to assess brain structure and neurochemistry before and six months after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

Obese Group

* Undergoing VSG-type bariatric surgery
* BMI > 30
* Current weight less than 400 lbs

Non-Obese Group

* Age 30-50
* BMI < 25

Exclusion Criteria:

Both Groups

* History of type 1 or type 2 diabetes
* History of stroke
* History of epilepsy
* History of Neurosurgical procedures
* Past or current history of severe psychiatric illness
* Pass or current history of alcohol or substance abuse
* Absence of metallic substances in body or ability to remove before imaging procedure
* History of claustrophobia or known inability to tolerate MRI
* Inability to consent

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Obese Group • Undergoing VSG-type bariatric surgery
  Non-Obese Group-healthy controls
  • BMI < 25
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Change insulin resistance and inflammatory markers | at baseline (before surgery) and 6 months post surgery
  Change in insulin resistance and blood inflammatory markers from baseline (before surgery) and at 6 months post surgery

SECONDARY OUTCOMES:
change in neurocognitive function testing | at baseline (before surgery) and 6 months post surgery
  changes in neurocognitive function testing from baseline (before surgery) and at 6 months post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Amir Moheet, Principal Investigator — University of Minnesota
Locations (1):
- Clinical and Translational Science Institute and Center for Magnetic Resonance Research, University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No